CLINICAL TRIAL: NCT03084393
Title: Postoperative Cognitive Dysfunction: Correlations With the Gene Polymorphism and the Concentrations of Plasma Homocysteine, Folic Acid and Vitamin B12.
Brief Title: POCD: Correlations With the Gene Polymorphism and the Concentrations of Plasma Homocysteine, Folic Acid and Vitamin B12.
Status: Completed | Type: Observational
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Han Yuan, Doctor-in-charge of Anesthetist, Xuzhou Medical University
Other Study IDs: XYFY2017-KL004-01
Record Dates: First submitted 2017-03-14; First posted 2017-03-20 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: non-cardiac surgery; Postoperative Cognitive Dysfunction
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: 215 Male and female patients undergoing non-cardiac surgery at the Affiliated Hospital of Xuzhou Medical University [Jiangsu China]. The investigators do the Mini-Mental score examination (MMSE) and neuropsychological tests 1 day before (baseline) and 1 week after surgery without safety issue. Patients will be divided into POCD and non-POCD groups according to the two times tests.
- non-surgical group: The investigators enroll 30 healthy volunteers and do the Mini-Mental score examination (MMSE) and neuropsychological tests at 1 day (baseline) and1 week without safety issue. The exclusive purpose of the non-surgical group is to aid in the POCD calculation according to the ISPOCD 1 study definition.

SUMMARY:
To study on the Postoperative Cognitive Dysfunction: Correlations With the Gene Polymorphism and the Concentrations of Plasma Homocysteine, Folic Acid and Vitamin B12. To explore whether the gene polymorphism and the concentrations of plasma homocysteine, folic acid and vitamin B12 could be used as predictor(s) of POCD and to provide reference for POCD prevention, early detection and timely diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Non-cardiac surgery patients;
* Age is greater than or equal to 60 years old;
* Han Nationality, mother tongue is chinese;
* The MMSE score: Illiteracy is greater than or equal to 17 points, primary school is greater than or equal to 20 points, higher secondary school is more than 24 points;
* The Geriatric Depression Scale (GDS) grade 1 or 2;
* The important function without serious heart, brain, liver, kidney, lung and other organs;
* The ASA class I or II;
* The people signed informed consent.

Exclusion Criteria:

* The diagnosis of neurological and psychiatric disorders, such as Alzheimer's disease, Parkinson's syndrome, multiple sclerosis, schizophrenia, depression, etc.;
* Had severe head and face disease, trauma history or history of surgery;
* The serious body disease and tobacco, wine and other substance abuse history;
* The presence of malignant tumor with shorter survival disease.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators included 215 Male and female patients undergoing non-cardiac surgery and 30 healthy volunteers at the affiliated hospital of Xuzhou Medical University.
Sampling Method: Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
the neuropsychological tests | 1 day before surgery(baseline)
  the neuropsychological tests to measure cognitive function, including the Trail Making Test, the Grooved Pegboard Test, the Digit Span Test, the Number-Symbol Replacement Test,the Finger Tapping Test, the Word Fluency Test and the Building Block Test.
Mini-Mental score examination [MMSE] | 1 day before surgery(baseline)
  Mini-Mental score examination [MMSE] used for screening of dementia
the neuropsychological tests | within the first 7 days (plus or minus 2 days) after surgery
  the neuropsychological tests to measure cognitive function, including the Trail Making Test, the Grooved Pegboard Test, the Digit Span Test, the Number-Symbol Replacement,the Test Finger Tapping Test, the Word Fluency Test and the Building Block Test.
Mini-Mental score examination [MMSE] | within the first 7 days (plus or minus 2 days) after surgery
  Mini-Mental score examination [MMSE] used for screening of dementia

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesia of the Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
within six months after the trial complete

REFERENCES:
- [Derived] Zhang ZF, Sun QC, Xu YF, Ding K, Dong MM, Han L, Abdul-Mannan, Han Y, Cao JL. Association between preoperative serum homocysteine and delayed neurocognitive recovery after non-cardiac surgery in elderly patients: a prospective observational study. Perioper Med (Lond). 2021 Nov 8;10(1):37. doi: 10.1186/s13741-021-00208-1. PMID 34743734